CLINICAL TRIAL: NCT05787249
Title: Improving Utilization of Supplemental Breast MRI Screening for Women With Extremely Dense Breasts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: UPCC 03123; P50CA244690 (NIH); 852666 (Registry Identifier: University of Pennsylvania Institutional Review Board)
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Breast density; Mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual care (no nudge) (No Intervention): Usual standard of care, no nudging.
- Provider nudge only (Experimental): Nudge sent to provider through EHR.
  Interventions: Behavioral: Provider nudge
- Patient nudge only (Experimental): Nudge sent to the patient through text messaging.
  Interventions: Behavioral: Patient nudge
- Patient and provider nudge (Experimental): Nudge sent to both provider through EHR, and to patient through text messaging.
  Interventions: Behavioral: Patient nudge; Behavioral: Provider nudge

INTERVENTIONS:
Behavioral: Patient nudge — Nudge directed to the patient with the aim of increasing the uptake of MRI in patients with extremely dense breasts
  Arms: Patient and provider nudge; Patient nudge only
Behavioral: Provider nudge — Nudge directed to the provider with the aim of increasing ordering of MRI in patients with extremely dense breasts
  Arms: Patient and provider nudge; Provider nudge only

SUMMARY:
The goal of this study is to increase MRI utilization among women with extremely dense breasts. The main question it seeks to answer is whether nudging of the provider, patient, or both increases the uptake of MRI among this group, and whether this effect differs between Black and White women.

DETAILED DESCRIPTION:
Women with dense breasts have 3-5-fold increased risk for breast cancer as women without dense breasts. Dense breast tissue can "mask" small tumors, leading to reduced mammography sensitivity. Recent randomized controlled trials demonstrate that supplemental breast MRI screening improves detection of small, invasive cancers that are not detected by mammography. In January 2022, a Pennsylvania law went into effect mandating insurance coverage of supplemental screening for women with extremely dense breasts. Currently only a small fraction of eligible women with extremely dense breasts are receiving supplemental breast MRI screening. Clinical pathways to identify patients who are eligible for insurance coverage of supplemental breast MRI screening and communicate this option to patients and providers are needed to ensure equitable access to supplemental screening. This study therefore proposes a stepped wedge cluster randomized clinical trial to determine whether electronic health record (EHR) and secure text message nudges increase utilization of supplemental breast MRI screening among eligible women with extremely dense breasts.

ELIGIBILITY:
Patient participants:

Inclusion Criteria:

* Women aged 40-74
* Recent non-actionable mammogram of less than 6 months
* Mammogram performed at Penn Center for Advanced Medicine, Penn Presbyterian Hospital, Pennsylvania Hospital, or Radnor
* Valid mobile phone number

Exclusion Criteria:

* Prior history of breast cancer
* No breast MRI within the past 2 years
* No prior actionable mammogram within 6 months
* No recent or concurrent ultrasound

Provider participants:

Inclusion Criteria:

* Provider needs to have ordered the initial screening mammogram
* Employed by Penn Health System and access to Penn Chart

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1358 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Ordering and/or scheduling of supplemental breast MRI | 6 months
  Whether a breast MRI is ordered and/or scheduled within 6 months of receiving a nudge.

SECONDARY OUTCOMES:
Ordering of breast MRI | 6 months
  Whether an MRI is ordered within 6 months of receiving a nudge. Analyzed separately from scheduling.
Scheduling of breast MRI | 6 months
  Whether an MRI is scheduled within 6 months of receiving a nudge. Analyzed separately from ordering.
Completion of breast MRI | 6 months
  Whether an MRI is completed within 6 months of receiving a nudge
False-positive rate | 6 months
  False-positive rate among those women who schedule and undergo MRI
Cancer detection rate | 6 months
  Cancer detection rate among those women who schedule and undergo MRI

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie McCarthy, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Bala-Cynwyd, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pettersson A, Graff RE, Ursin G, Santos Silva ID, McCormack V, Baglietto L, Vachon C, Bakker MF, Giles GG, Chia KS, Czene K, Eriksson L, Hall P, Hartman M, Warren RM, Hislop G, Chiarelli AM, Hopper JL, Krishnan K, Li J, Li Q, Pagano I, Rosner BA, Wong CS, Scott C, Stone J, Maskarinec G, Boyd NF, van Gils CH, Tamimi RM. Mammographic density phenotypes and risk of breast cancer: a meta-analysis. J Natl Cancer Inst. 2014 May 10;106(5):dju078. doi: 10.1093/jnci/dju078. PMID 24816206
- [Background] Bond-Smith D, Stone J. Methodological Challenges and Updated Findings from a Meta-analysis of the Association between Mammographic Density and Breast Cancer. Cancer Epidemiol Biomarkers Prev. 2019 Jan;28(1):22-31. doi: 10.1158/1055-9965.EPI-17-1175. Epub 2018 Sep 11. PMID 30206060
- [Background] Comstock CE, Gatsonis C, Newstead GM, Snyder BS, Gareen IF, Bergin JT, Rahbar H, Sung JS, Jacobs C, Harvey JA, Nicholson MH, Ward RC, Holt J, Prather A, Miller KD, Schnall MD, Kuhl CK. Comparison of Abbreviated Breast MRI vs Digital Breast Tomosynthesis for Breast Cancer Detection Among Women With Dense Breasts Undergoing Screening. JAMA. 2020 Feb 25;323(8):746-756. doi: 10.1001/jama.2020.0572. PMID 32096852
- [Background] Veenhuizen SGA, de Lange SV, Bakker MF, Pijnappel RM, Mann RM, Monninkhof EM, Emaus MJ, de Koekkoek-Doll PK, Bisschops RHC, Lobbes MBI, de Jong MDF, Duvivier KM, Veltman J, Karssemeijer N, de Koning HJ, van Diest PJ, Mali WPTM, van den Bosch MAAJ, van Gils CH, Veldhuis WB; DENSE Trial Study Group. Supplemental Breast MRI for Women with Extremely Dense Breasts: Results of the Second Screening Round of the DENSE Trial. Radiology. 2021 May;299(2):278-286. doi: 10.1148/radiol.2021203633. Epub 2021 Mar 16. PMID 33724062
- [Background] Weinstein SP, Korhonen K, Cirelli C, Schnall MD, McDonald ES, Pantel AR, Zuckerman S, Borthakur A, Conant EF. Abbreviated Breast Magnetic Resonance Imaging for Supplemental Screening of Women With Dense Breasts and Average Risk. J Clin Oncol. 2020 Nov 20;38(33):3874-3882. doi: 10.1200/JCO.19.02198. Epub 2020 Sep 15. PMID 32931396
- [Background] Expert Panel on Breast Imaging; Weinstein SP, Slanetz PJ, Lewin AA, Battaglia T, Chagpar AB, Dayaratna S, Dibble EH, Goel MS, Hayward JH, Kubicky CD, Le-Petross HT, Newell MS, Sanford MF, Scheel JR, Vincoff NS, Yao K, Moy L. ACR Appropriateness Criteria(R) Supplemental Breast Cancer Screening Based on Breast Density. J Am Coll Radiol. 2021 Nov;18(11S):S456-S473. doi: 10.1016/j.jacr.2021.09.002. PMID 34794600
- [Background] Wolf, Tom. "Insurance Company Law of 1921 - Coverage for Mammographic Examinations." The Office Website for the Pennsylvania General Assembly, Pennsylvania General Assembly, 2020, https://www.legis.state.pa.us/cfdocs/legis/li/uconsCheck.cfm?yr=2020&sessInd=0&act=52.
- [Background] Niraula S, Biswanger N, Hu P, Lambert P, Decker K. Incidence, Characteristics, and Outcomes of Interval Breast Cancers Compared With Screening-Detected Breast Cancers. JAMA Netw Open. 2020 Sep 1;3(9):e2018179. doi: 10.1001/jamanetworkopen.2020.18179. PMID 32975573
- [Background] Monsees BS. The Mammography Quality Standards Act. An overview of the regulations and guidance. Radiol Clin North Am. 2000 Jul;38(4):759-72. doi: 10.1016/s0033-8389(05)70199-8. PMID 10943276
- [Background] Sedrak MS, Myers JS, Small DS, Nachamkin I, Ziemba JB, Murray D, Kurtzman GW, Zhu J, Wang W, Mincarelli D, Danoski D, Wells BP, Berns JS, Brennan PJ, Hanson CW, Dine CJ, Patel MS. Effect of a Price Transparency Intervention in the Electronic Health Record on Clinician Ordering of Inpatient Laboratory Tests: The PRICE Randomized Clinical Trial. JAMA Intern Med. 2017 Jul 1;177(7):939-945. doi: 10.1001/jamainternmed.2017.1144. PMID 28430829
- [Background] Patel MS, Kurtzman GW, Kannan S, Small DS, Morris A, Honeywell S Jr, Leri D, Rareshide CAL, Day SC, Mahoney KB, Volpp KG, Asch DA. Effect of an Automated Patient Dashboard Using Active Choice and Peer Comparison Performance Feedback to Physicians on Statin Prescribing: The PRESCRIBE Cluster Randomized Clinical Trial. JAMA Netw Open. 2018 Jul 6;1(3):e180818. doi: 10.1001/jamanetworkopen.2018.0818. PMID 30646039
- [Background] Takvorian SU, Bekelman J, Beidas RS, Schnoll R, Clifton ABW, Salam T, Gabriel P, Wileyto EP, Scott CA, Asch DA, Buttenheim AM, Rendle KA, Chaiyachati K, Shelton RC, Ware S, Chivers C, Schuchter LM, Kumar P, Shulman LN, O'Connor N, Lieberman A, Zentgraf K, Parikh RB. Behavioral economic implementation strategies to improve serious illness communication between clinicians and high-risk patients with cancer: protocol for a cluster randomized pragmatic trial. Implement Sci. 2021 Sep 25;16(1):90. doi: 10.1186/s13012-021-01156-6. PMID 34563227
- [Background] Jenssen BP, Schnoll R, Beidas R, Bekelman J, Bauer AM, Scott C, Evers-Casey S, Nicoloso J, Gabriel P, Asch DA, Buttenheim A, Chen J, Melo J, Shulman LN, Clifton ABW, Lieberman A, Salam T, Zentgraf K, Rendle KA, Chaiyachati K, Shelton R, Wileyto EP, Ware S, Leone F. Rationale and protocol for a cluster randomized pragmatic clinical trial testing behavioral economic implementation strategies to improve tobacco treatment rates for cancer patients who smoke. Implement Sci. 2021 Jul 15;16(1):72. doi: 10.1186/s13012-021-01139-7. PMID 34266468
- [Derived] McCarthy AM, Fernandez Perez C, Beidas RS, Bekelman JE, Blumenthal D, Mack E, Bauer AM, Ehsan S, Conant EF, Wheeler BC, Guerra CE, Nunes LW, Gabriel P, Doucette A, Wileyto EP, Buttenheim AM, Asch DA, Rendle KA, Shelton RC, Fayanju OM, Ware S, Plag M, Hyland S, Gionta T, Shulman LN, Schnoll R. Protocol for a pragmatic stepped wedge cluster randomized clinical trial testing behavioral economic implementation strategies to increase supplemental breast MRI screening among patients with extremely dense breasts. Implement Sci. 2023 Nov 24;18(1):65. doi: 10.1186/s13012-023-01323-x. PMID 38001506